CLINICAL TRIAL: NCT01098344
Title: A Cancer Research UK Phase I Trial of an Oral Notch Inhibitor (MK-0752) in Combination With Gemcitabine in Patients With Stage III and IV Pancreatic Cancer
Brief Title: MK0752 and Gemcitabine Hydrochloride in Treating Patients With Stage III and IV Pancreatic Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000669535; CRUK-CR0720-11; CRUK-MK-0752; EUDRACT-2008-004829-42
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; stage IV pancreatic cancer; duct cell adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 3-(4-((4-chlorophenyl)sulfonyl)-4-(2,5-difluorophenyl)cyclohexyl)propanoic acid; Gemcitabine

INTERVENTIONS:
Drug: Notch signaling pathway inhibitor MK0752
Drug: gemcitabine hydrochloride
Other: imaging biomarker analysis
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: MK0752 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving MK0752 together with gemcitabine hydrochloride may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of giving MK0752 together with gemcitabine hydrochloride and to see how well it works in treating patients with stage III or IV pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the recommended phase II dose of MK0752 in combination with gemcitabine hydrochloride in patients with unresectable stage III and IV pancreatic cancer. (Phase I)

Secondary

* To evaluate tumor response in patients treated with this regimen.
* To determine the time to disease progression and 6 months and 1-year survival.
* To determine the percentage of change in CA19-9 levels.

Tertiary

* To assess target inhibition of MK0752 in plasma.
* To explore the feasibility of measuring MK0752 levels in tumor tissue.
* To establish relationships between measures of tumor expression of molecular target and objective tumor response.
* To determine the pharmacokinetic profile of MK0752 in plasma when administered with and without gemcitabine hydrochloride.

OUTLINE: This is a multicenter, phase I, dose-escalation study of MK0752 and gemcitabine hydrochloride.

Patients receive gemcitabine hydrochloride IV on days 1, 8, and 15. Patients receive oral MK0752 on days -14, -7, 1, 8, 15, and 22 in course 1 only and on days 1, 8, 15, and 22 beginning in course 2 and for all subsequent courses. Treatment with MK0752 and gemcitabine hydrochloride repeats every 28 days* for 6 courses in the absence of disease progression or unacceptable toxicity.

NOTE: *The first course is 42 days.

Patients undergo biopsy of tumor at baseline and on day -7. Tumor samples are analyzed to determine Notch pathway inhibition via IHC and qualitative RT-PCR analysis and for MK0752 concentrations. Hair follicle (from the head) samples are collected at baseline and on day -7 to determine Notch pathway inhibition via RT-PCR. Blood samples are collected periodically to determine changes in CA 19-9 levels and MK0752 concentrations.

After completion of study treatment, patients are followed for 28 days and then every 2 months for 1 year. Patients will then be followed up as part of their normal clinic visits for up to one year after the last patient was treated on the study.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed ductal adenocarcinoma of the pancreas

  * Stage III and IV, unresectable disease
* Assessable disease by endoscopic ultrasound or CT guidance
* Tissue that is assessed by the Investigator as being accessible to biopsy - for patients recruited to dose escalation phase where three previous patients have not already provided biopsies
* No known brain metastases

  * Patients with stable symptoms within the past 4 weeks, on a stable dose of steroids, and able to give informed consent are eligible

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Life expectancy ≥ 12 weeks
* Hemoglobin ≥ 9.0 g/dL
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 2.5 times ULN (≤ 5 times ULN if due to liver metastases)
* PT ≤ 1.5 times ULN
* Creatinine clearance ≥ 50 mL/min (uncorrected)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use two forms of highly effective contraception (females) 4 weeks prior to, during, and for 6 months after completion of study therapy or 1 form of highly effective contraception (males) during and for 6 months after completion of study therapy
* Written (signed and dated) informed consent and capable of cooperating with treatment and follow-up
* No nonmalignant systemic disease, including active uncontrolled infection, that confers a high medical risk to the patient
* No known serologically positive HIV or hepatitis B or C infection
* No other concurrent malignancies except adequately treated cone-biopsied carcinoma in situ of the uterine cervix, basal or squamous cell carcinoma of the skin, or cancer survivors who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease ≥ 5 years, and are deemed at negligible risk for recurrence
* No concurrent congestive heart failure
* No prior history of cardiac disease (New York Heart Association class III-IV disease), cardiac ischemia, or cardiac arrhythmia
* No other condition that, in the investigator's opinion, would not make the patient a good recommendation for the clinical trial

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior treatments
* Previous chemotherapy for advanced disease is permitted. If gemcitabine treatment was given previously, the patient must have tolerated a dose of at least 800mg/m2. Previous chemotherapy for malignant disease must be complete at least 3 weeks before treatment on this trial (six weeks for mitomycin C)
* No major thoracic or abdominal surgery from which the patient has not yet recovered
* No concurrent participation or planned participation in another interventional clinical study

  * Concurrent participation in an observational study allowed
* No concurrent warfarin

  * Low molecular weight heparin allowed
* No concurrent radiotherapy (except palliative for bone pain), endocrine therapy, or immunotherapy
* No other concurrent anticancer therapy or investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose of MK0752 in combination with gemcitabine hydrochloride OR the single agent recommended Phase II dose in combination with either 800 mg/m² or 1000 mg/m² as agreed by DDO and clinicians
Adverse event and severity according to NCI CTCAE Version 4.02

SECONDARY OUTCOMES:
Complete response, partial response, or stable disease as defined by RECIST criteria
Progression-free survival
Survival at 1 year
Percentage change in CA19-9 levels
Plasma concentrations of MK0752

CONTACTS AND LOCATIONS:
Overall Officials: Duncan Jodrell, MD, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - Addenbrooke's Hospital, Cambridge, England
  - Leicester Royal Infirmary, Leicester, England
  - Barts and the London School of Medicine, London, England
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - St James' Hospital, Leeds